CLINICAL TRIAL: NCT02964546
Title: Impact of the Choice of Glomerular Filtration Rate-Estimating Equations on Plasmatic Concentrations of Direct Oral Anticoagulants in Elderly Patients With Atrial Fibrillation
Brief Title: Glomerular Filtration Rate-Estimating Equations During Use of Direct Oral Anticoagulants in Elderly Patients
Acronym: REINACO
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9539; 2015-A00453-46 (Other: FRANCE: Agence Nationale de Sécurité du Médicament et des Produits de santé)
Record Dates: First submitted 2016-09-09; First posted 2016-11-16 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation; Elderly Patients; Chronic Kidney Disease
Keywords: direct oral anticoagulants; atrial fibrillation; renal function; ckd-epi; plasmatic concentration
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood sample
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 2 additional tubes of blood samples are collected during a blood sample realized for the patient's care

SUMMARY:
Atrial fibrillation in the elderly is a complex condition due to the high number of frequently associated comorbidities such kidney disease. Direct oral anticoagulants (dabigatran, rivaroxaban and apixaban) are indicated for preventing thromboembolic events but renal function should be closely monitored for this age group when these drugs are used. Dosing recommendations for prevention of stroke are based on renal clearance of creatinine (ClCr) estimated using the Cockcroft-Gault formula. It is well known that ClCr estimates predict a steeper decline with advancing age than Glomerular Filtration Rate (GFR) estimates. This raises the possibility that substitution of commonly reported GFR for estimated CrCl could result in different plasmatic concentrations of oral direct anticoagulants. The aim of this study was to compare estimates of ClCr and GFR and determine the impact on the plasmatic concentration of these drugs in elderly patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

Patients with non-valvular atrial fibrillation -treated with dabigatran, rivaroxaban or apixaban - patients affiliated to national social health system -patients who agreed to ethical concerns of the study

Exclusion Criteria:

Patients with consultation or hospitalization that made impossible a veinous punction at the steady state residual concentration time -Patients under guardianship or trusteeship

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with non-valvular atrial fibrillation treated with dabigatran, rivaroxaban or apixaban
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
renal function estimated by different glomerular filtration rate equations and by clearance of creatinine formula | At the inclusion

SECONDARY OUTCOMES:
plasmatic activity of direct oral anticoagulant at steady state residual time (anti-Xa or anti-IIa) | At the inclusion
plasmatic concentration of direct oral anticoagulant at steady state residual time | At the inclusion
Number of haemorrhagic or thrombotic adverse events (serious or not) affecting patients | At 1 month
  Reported by a trained physician after a phone interview with the patient coupled with medication adherence assessment using 6-item Moriksy scale. An internal questionnaire will be used to collect data.
Number of haemorrhagic or thrombotic adverse events (serious or not) and unexpected events affecting patients | At 6 months
  Reported by a trained physician after a phone interview with the general practitioner and the patient coupled with medication adherence assessment using 6-item Moriksy scale. An internal questionnaire will be used to collect data.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No